CLINICAL TRIAL: NCT00423722
Title: Parenteral Hydration in Advanced Cancer Patients - A Randomized Controlled Trial
Brief Title: Parenteral Hydration in Advanced Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2006-0494; R01CA122292-01 (NIH); NCI-2010-00984 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Results first posted 2015-12-17 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Advanced Cancer; Dehydration
Keywords: Advanced Cancer; Hospice Care; Caregiver; Saline; Hydration; Dehydration
MeSH Terms: conditions — Dehydration | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydration: Normal Saline (salt water) (Experimental): Group 1: 1,000 ml of normal saline (0.9% sodium chloride) parenterally over 4 hours daily
  Interventions: Drug: Saline
- Placebo: Lower Saline (Placebo Comparator): Group 2: Lower Amount of Normal Saline (salt water); 100 ml of normal saline (0.9% sodium chloride) parenterally over 4 hours daily.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Saline — 1,000 ml of normal saline (0.9% sodium chloride) parenterally over 4 hours daily.
  Arms: Hydration: Normal Saline (salt water)
Drug: Saline — 100 ml of normal saline (0.9% sodium chloride) parenterally over 4 hours daily.
  Arms: Placebo: Lower Saline

SUMMARY:
The goal of this clinical research study is to learn whether being hydrated (given liquids) through a catheter in a vein or in the tissue under the skin can improve symptoms of dehydration.

Objectives:

1.1 Determine whether parenteral hydration is superior to placebo in improving symptoms associated with dehydration (such as fatigue, myoclonus, sedation, and hallucinations) in advanced cancer patients receiving hospice care.

1.2 Determine whether parenteral hydration is superior to placebo in delaying the onset or reducing the severity of delirium in patients with advanced cancer receiving hospice care.

1.3 Describe the meaning patients and primary caregivers attribute to dehydration and re-hydration at the end of patient's lives.

DETAILED DESCRIPTION:
For Caregivers:

Symptoms of dehydration may include fatigue, muscle contractions, the need for sedation (calming medication), and hallucinations (where something is sensed that is not actually there). Hydration allows the body to get rid of the waste products from medications and other chemicals. When the fluid levels in the body are increased, the brain function may directly improve.

If the patient under your care is found to be eligible to take part in this study, he or she will be randomly assigned (as in the toss of the coin) to one of 2 groups. Participants in Group 1 will receive normal saline (salt water) once a day. Participants in Group 2 will receive a lower amount of normal saline once a day. This lower amount is small enough to be considered a placebo. Doctors call something a placebo if it looks like the substance being tested but has no active ingredients (or in this case, few active ingredients).

Both you and the patient will be asked to complete a number of questionnaires at the beginning of the study, on Days 1-7, and then every 3-5 days after that. Your questionnaires will ask about the feelings you may have about hydration and the care that you are providing to the patient. Each day's questionnaires will take about 30 minutes.

Both you and the patient will also be interviewed by researchers at the beginning of the study and on Day 4 (+/- 2 days). The interviews will include questions about what it has been like for the patient to get fluids, whether the fluid was more like food or medicine, whether the patient has ever gotten dehydrated, and how you manage the patient's care. The interviews should each take about 30 minutes. The interviews in this study will be audio taped so the information can be studied by researchers. Only the research staff will listen to the audio tape of the interviews.

If the patient goes off study, your participation in the study will be over.

This is an investigational study. Up to 150 patients and 150 caregivers will take part in this study. All will be enrolled at M. D. Anderson.

For Patients:

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. You will be asked to complete a questionnaire. It will ask questions about your cancer diagnoses, the medications you are taking, and the symptoms you are having. The questionnaire also asks about your memory of being dehydrated, what it was like for you to get fluids, how you manage your care, and whether the fluid was more like food or medicine. It should take about 30 minutes to complete.

Both you and your caregiver will also be interviewed by researchers. There will be questions about what it has been like for you to get fluids, whether the fluid was more like food or medicine, and whether you have ever gotten dehydrated. Each interview should take about 30 minutes. The interviews in this study will be audio taped so the information can be studied by researchers.

The study staff will also check you for symptoms of muscle contraction, one of the signs of dehydration. The study staff will videotape your face, arms, hands, legs and toes for a total 3-5 minutes on Days 1, 4, and 7, and then every 3-5 days after that.

As part of the screening tests, you will also have blood drawn (about 2 teaspoons) for routine tests. You will be asked questions about your ability to perform daily activities (performance status evaluation). You will be asked about any side effects you may have, including muscle contractions. You will also be asked to list any pain medications or other medications that you take.

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of the coin) to one of two groups. Participants in Group 1 will receive normal saline (salt water) once a day. Participants in Group 2 will receive a lower amount of normal saline once a day. This lower amount is small enough to be considered a placebo. Doctors call something a placebo if it looks like the substance being tested but has no active ingredients (or in this case, few active ingredients). You will have an equal chance of being placed in either group. Neither you nor any of the medical staff or researchers on this study will know which dose you are receiving.

The research nurse will ask you to complete several questionnaires that ask questions about dehydration and the symptoms you may have experienced, including fatigue. The questionnaires will be completed on Days 1-7, and then every 3-5 days after that. In total, each day's questionnaires should take about 30 minutes. Your caregiver will also be asked about his or her memory of your dehydration. On Day 7, you will have blood drawn (about 2 teaspoons) for routine tests.

Both you and your caregiver will also be interviewed by researchers on Day 4 (+/- 2 days), and then every 3-5 days after that. The interviews will be like the ones at screening.

Starting on Day 1 of the study, you will receive saline through a catheter in a vein (over 4 hours) every day. If you already have a central venous catheter, you will receive the saline through that catheter. If you do not have a central venous catheter, the saline will be infused under the skin. Either way, the infusion will last about 4 hours.

During each infusion, an infusion research nurse will check to make sure that the saline is given properly. This nurse will know which treatment group you have been assigned to.

Every day, the research nurse will ask you about the dehydration and any side effects you may have. Every day, the research nurse will also check the place where the infusion is given to make sure there is no infection.

On Days 1-7 and then every 3-5 days, the research nurse will also check for any dehydration symptoms including the need for sedation, any restless feelings or actions, and/or muscle contractions. You will have a performance status evaluation daily. On Days 1-7, the research nurse will ask about any pain medications or other medications that you have taken.

Every day, 2 hours [+/- 3 hours] after the infusion ends, you will also be checked by an assessment research nurse who will not know which treatment group you are in. The assessment research nurse will ask about any symptoms you may have. The study staff will also check you for symptoms of muscle contraction, one of the signs of dehydration. The study staff will videotape your face, arms, hands, legs and toes for a total 3-5 minutes on Days 1, 4, and 7, and then every 3-5 days after that.

You may remain on study to receive the daily infusions for as long as you are benefitting up to Day 14 [+/- 3 days]. On Day 14 [+/- 3 days] you will be taken off study, and you will have off study assessments, which include questions about your symptoms including fatigue, performance status, medications you are taking, and dehydration symptoms. If intolerable side effects occur, you will be taken off study and given appropriate medical care. If you wish to continue receiving hydration fluids after you are taken off study [Day 14 +/- 3 days], you may discuss this option with your attending hospice physician. You may receive a liter of normal saline each day under the skin. Treatment will be given by hospice nurse. Fluid will be provided to you free of charge.

This is an investigational study. Up to 150 patients and 150 caregivers will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced cancer (local recurrence or metastatic disease) admitted to hospice care
2. Patients have reduced oral intake of fluids, as determined by clinical assessment.
3. Patients exhibit evidence of mild or moderate dehydration as defined by decreased skin turgor in subclavicular region (more than 2 seconds), plus a score of >/= 2/5 in the clinical dehydration assessment
4. In addition to fatigue, (expected to be present in all patients based on our pilot study), patients must score >/= 1 on a 0 to 10 scale (0=no symptom, 10= the worst possible symptom) of two of the three other target symptoms (hallucinations, sedation, and myoclonus) scored
5. Patients are 18 years of age or older
6. Patients have life expectancy of >/= 1 week as determined by their treating physicians
7. Patients who score < 13 (normal range) in the Memorial Delirium Assessment Scale (MDAS) and are able to give written informed consent
8. Patients must be able to tolerate the parenteral treatment application device (butterfly cannula or intravenous access)
9. Patients must have a primary caregiver
10. Patients must reside within 60 miles of M. D. Anderson Cancer Center. Exception to this is for patients referred from Odyssey Health Care of Conroe, patients referred from this site must reside within 75 miles of M.D. Anderson Cancer Center.
11. Inclusion criteria of family caregivers: The family caregiver is a person who is patient's spouse, parent, sibling. child or significant other
12. The family caregiver must reside with the patient and is responsible for the care of the patient. Exception to this is for patients who are admitted to In Patient hospice or nursing homes/rehabilitation centers and are under the care of the hospice.
13. The family caregiver must be 18 years of age or older
14. The family caregiver must be willing to be interviewed by the research nurse and sign written informed consent

Exclusion Criteria:

1. Patient's refuse to participate in the study or are not competent to give informed consent
2. Patients are suffering from severe dehydration defined as decreased blood pressure or low perfusion of limbs, decreased level of consciousness, or no urine output for 12 hours
3. Patients with history or clinical evidence of renal failure. Creatinine >1.5 x *Upper Limit of Normal. (M.D. Anderson Cr ULN=1.5 mg/dl). Therefore, a patient with Creatinine of (CR)> 2.25 mg/dl will be excluded.
4. Patients with history or clinical evidence of congestive heart failure
5. Patients who are not able to complete the baseline assessment forms
6. Patients have history of bleeding disorders demonstrated by clinical evidence of active bleeding, hematuria, hematoma, ecchymoses, and petechiae
7. Patients with brain metastasis, leptomeningeal disease or primary brain tumors will be eligible for participation in this study as long as there is no evidence of altered mental status as demonstrated by a normal score on the Memorial Delirium Assessment Scale (MDAS).
8. The family caregiver refuses to participate in the study
9. The family caregiver has difficulty understanding the intent of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2007-01-09 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Bruera, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (5):
  - Odyssey Healthcare of Conroe, Conroe, Texas
  - Houston Hospice and Palliative Care System, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Odyssey Healthcare of Houston, Houston, Texas
  - Vitas Healthcare, Houston, Texas

REFERENCES:
- [Result] Bruera E, Hui D, Dalal S, Torres-Vigil I, Trumble J, Roosth J, Krauter S, Strickland C, Unger K, Palmer JL, Allo J, Frisbee-Hume S, Tarleton K. Parenteral hydration in patients with advanced cancer: a multicenter, double-blind, placebo-controlled randomized trial. J Clin Oncol. 2013 Jan 1;31(1):111-8. doi: 10.1200/JCO.2012.44.6518. Epub 2012 Nov 19. PMID 23169523
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 01/07/2007 - 05/02/2011. Participating sites included Silverado Hospice, Odyssey Hospice, Vitas Hospice, Houston Hospice and Christus Visiting Nurse Association (VNA) Hospice in the Greater Houston area.
Period: Overall Study
Arm/Group | Hydration: Normal Saline (Salt Water) | Placebo: Lower Saline
Started | 63 | 66
Completed | 49 | 53
Not Completed | 14 | 13
Not completed — Death | 4 | 4
Not completed — Declined to participate | 2 | 3
Not completed — Unable to complete questionnaires | 4 | 4
Not completed — Withdrawal by Subject | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydration: Normal Saline (Salt Water) | Placebo: Lower Saline | Total
Number analyzed (Participants) | 63 | 66 | 129
Age, Continuous [Mean (Full Range); unit: years] | 67 [43 to 92] | 67 [41 to 92] | 67 [41 to 92]
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 29 | 56
  >=65 years | 36 | 37 | 73
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 36 | 61
  Male | 38 | 30 | 68
Region of Enrollment [Number; unit: participants]
  United States | 63 | 66 | 129

OUTCOME MEASURES:

1. Primary Outcome: Participant Reduced Symptom Burden
Description: Symptom burden, assessed using the Edmonton Symptom assessment scale, which has been validated in the cancer population. Participants are asked to rate the severity of their symptoms over the previous 24 hours using a numerical rating scale of 0-10, with 0 meaning that the symptom is absent and 10 meaning the worst possible symptom. The mean is a composite outcome where change in the sum of 4 dehydration symptoms (fatigue, myoclonus, sedation and hallucinations) between day 4 and baseline ranged from 0-40 daily. The reported value was the mean of average change in patients' scores per group.
Time Frame: From Baseline to 4 Days Later (Daily assessments at 2 hours [+/- 3 hours] after the completion of 4-Hour infusion)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Hydration: 1,000 ml of normal saline (0.9% sodium chloride) parenterally over 4 hours daily.
- Placebo: Lower Amount of Normal Saline (salt water); 100 ml of normal saline (0.9% sodium chloride) parenterally over 4 hours daily.
Arm/Group | Hydration | Placebo
Number analyzed (Participants) | 49 | 53
units on a scale | -3.3 (7.6) | -2.8 (9.2)

2. Secondary Outcome: Reduced Symptom Burden as Measured by RASS, MDAS and UMRS
Description: Participants rated delirium, quality of life, and overall survival using Richmond agitation sedition scale (RASS) where +4 is "Combative" to -5 is "Unarousable"; Memorial delirium assessment scale (MDAS), a ten-item, clinician-rated scale from 0 (none) to 3 (severe) for severity of delirium, for a total range of 0-30; and Unified Myoclonus Rating Scale (UMRS) 5-functional scores rated 0 to 4, for a total range of 0-20 where higher scores indicate more severe involuntary movements. Higher scores indicate worse outcomes for each scale, i.e. RASS more agitation, MDAS more delirium and UMRS more severe involuntary movements. The mean represents change in combined participant daily scores for each scale between Baseline and Day 4 assessments then separately Day 7 assessments. Reported value is mean of average change in patients' scores per group. Reported values reflect changes from baseline, either median decreases (less than 0), no change (0) or increases (greater than 0).
Time Frame: Baseline to Day 7
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Hydration (Baseline and Day 4); Hydration (Baseline and Day 7): 1,000 ml of normal saline (0.9% sodium chloride) parenterally over 4 hours daily.
- Placebo (Baseline and Day 4); Placebo (Baseline and Day 7): Lower Amount of Normal Saline (salt water); 100 ml of normal saline (0.9% sodium chloride) parenterally over 4 hours daily.
Arm/Group | Hydration (Baseline and Day 4) | Placebo (Baseline and Day 4) | Hydration (Baseline and Day 7) | Placebo (Baseline and Day 7)
Number analyzed (Participants) | 49 | 53 | 49 | 53
units on a scale
  RASS | 0 [-1 to 0] | 0 [-2 to 0] | 0 [-1 to 0] | -1 [-2 to 0]
  MDAS | 1 [-2 to 5.8] | 3.5 [-0.3 to 14.5] | 2 [-2 to 10] | 2.5 [-1 to 14]
  UMRS | 0 [0 to 3] | 0 [0 to 8] | 1 [0 to 5.8] | 0 [0 to 5.5]

3. Secondary Outcome: Change in Quality of Life and Fatigue as Measured by FACIT-F and FACT-G From Baseline to Day 7
Description: Change between Day 7 to Baseline in FACIT-F (Functional Assessment of Chronic illness Therapy-Fatigue) & FACT-G (Functional Assessment of Cancer Therapy-General) scores. Participants rate quality of life using FACT-G consisting of 33 questions with 5 domains assessing physical and social, emotional & functional well being & relationship with physician, remaining 5 assess extent to which each domain affects overall quality of life on 5-point scale from 0 (not at all) to 4 (very much); total score obtained by summing individual subscale scores (0-132). FACIT-F consists of 13 items where participants rate intensity of fatigue & its related symptoms on a scale of 0-4 from 0 "not at all" to 4 "very much." The responses to FACIT fatigue questionnaire are each measured on 4-point Likert scale with total score ranges from 0 to 52. High scores represent less fatigue. Reported is the mean change of the summed value of all reported scores for the FACT-G or the FACIT-F from baseline to Day 7.
Time Frame: Baseline to Day 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hydration (Baseline and Day 7) | Placebo (Baseline and Day 7)
Number analyzed (Participants) | 44 | 49
units on a scale
  FACT-G | 6.7 (11.2) | 2.6 (16.7)
  FACIT-F | 9.1 (17.9) | 1.4 (25.6)

4. Secondary Outcome: Reduced Symptom Burden (From Baseline to 7 Days Post Infusion)
Description: Secondary outcomes included delirium, quality of life, and overall survival. The Nursing delirium screening scale (NuDESC) was used to assess delirium. NuDESC is a validated observational instrument conducted by research staff based on input from family caregivers. Five symptoms (disorientation, inappropriate behavior, inappropriate communication, illusions or hallucinations, and psychomotor retardation) are each given a score from 0 to 2, for a possible total score of 10. A higher NuDESC score indicates increased symptoms of delirium. It was observed a trend for lesser decline (delirium) in the hydration group, and significant worsening of night-time NuDESC scores in the placebo group.
Time Frame: Baseline to Day 7 (Daily assessments at 2 hours [+/- 3 hours] after the completion of 4-Hour infusion)
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Hydration (Baseline and Day 4) | Placebo (Baseline and Day 4) | Hydration (Baseline and Day 7) | Placebo (Baseline and Day 7)
Number analyzed (Participants) | 49 | 53 | 49 | 53
units on a scale
  NuDESC Day | 0 [-1 to 1] | 0 [-1 to 2] | 0 [0 to 0] | 0 [0 to 1]
  NuDESC Evening | 0 [-1 to 1] | 0 [-1 to 2] | 0 [-1 to 1] | 0 [-1 to 3]
  NuDESC Night | 0 [-1 to 0] | 0 [-1 to 2] | 0 [-1 to 1] | 0 [-1 to 1]

5. Secondary Outcome: Change in Dehydration as Measured by Dehydration Assessment Scale
Description: Dehydration was assessed by using the Dehydration Assessment Scale on the basis of three physical findings, moisture on the mucous membranes of the mouth (0=moist, 1=somewhat dry, 2=dry), axillary moisture (0=moist, 1=dry) and sunkenness of the eyes (0=normal, 1=slight sunken, 2=sunken). These signs are selected due to their significant correlations with biological dehydration, as previously confirmed by elderly patients. The dehydration score (range 0-7) is calculated as the total of these 3 scores, a higher score indicates a higher level of dehydration. The reported value was the mean of average change in patients' scores per group.
Time Frame: Baseline to Day 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hydration (Baseline and Day 4) | Placebo (Baseline and Day 4) | Hydration (Baseline and Day 7) | Placebo (Baseline and Day 7)
Number analyzed (Participants) | 49 | 53 | 49 | 53
units on a scale | -0.8 (1.5) | -0.6 (1.4) | -1.0 (1.7) | -0.5 (1.4)

ADVERSE EVENTS:
Time Frame: Adverse event reporting collected an average of 7 days, up to 10 days for participant study period from January 2007 to May 2011.
Groups:
- Hydration; Placebo: Change Between Day 4 and Baseline
Arm/Group | Hydration | Placebo
Serious Adverse Events (participants affected / at risk) | 18/63 | 13/66
Other Adverse Events (participants affected / at risk) | 42/63 | 48/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydration (N=63) | Placebo (N=66)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Bone pain (General disorders) | 1 (1) | 0 (0)
BUN Increase (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 4 (4) | 1 (1)
Involuntary Movement (Nervous system disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 2 (2) | 1 (1)
Psychosis (Psychiatric disorders) | 1 (1) | 1 (1)
Seizures (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 4 (4) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Calcium, Serum-high (Investigations) | 0 (0) | 1 (1)
Death NOS (General disorders) | 0 (0) | 1 (1)
Disease Progression NOS (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than .5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydration (N=63) | Placebo (N=66)
Anorexia (Metabolism and nutrition disorders) | 10 (11) | 4 (4)
Anxiety (Psychiatric disorders) | 5 (7) | 4 (6)
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
BUN increase (Blood and lymphatic system disorders) | 2 (2) | 6 (6)
Cardiac Arrhytmia (Cardiac disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 2 (3)
Constipation (Gastrointestinal disorders) | 5 (6) | 4 (5)
Creatine (Investigations) | 1 (2) | 1 (1)
Depression (Psychiatric disorders) | 8 (8) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 6 (9)
Dysuria (Infections and infestations) | 1 (1) | 2 (2)
Edema (General disorders) | 27 (151) | 25 (100)
Fatigue (General disorders) | 13 (17) | 12 (13)
Fever (General disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hemorrhage (General disorders) | 1 (1) | 0 (0)
Incontinence, Urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 2 (3) | 0 (0)
Involuntary Movement (Nervous system disorders) | 5 (14) | 7 (7)
Metabolic/laboratory (Investigations) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 2 (3)
Nausea (Gastrointestinal disorders) | 14 (18) | 9 (16)
Neuropathy: Sensory (Nervous system disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 11 (20) | 10 (19)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Psychosis (Psychiatric disorders) | 8 (12) | 7 (12)
Respiratory Symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 12 (20) | 15 (23)
Vomiting (Gastrointestinal disorders) | 4 (5) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Calcium-Serum high (Investigations) | 0 (0) | 2 (2)
Consciousness level depressed (Nervous system disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Earache (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hallucinations (Nervous system disorders) | 0 (0) | 1 (1)
Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (3)
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Jaundice (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neurology (Nervous system disorders) | 0 (0) | 1 (1)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Urine color change (Renal and urinary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study had a planned sample size of 150 participants but due to funding issues recruitment was halted after 129 patients; additionally, participants with delirium or severe dehydration were excluded for logistic purposes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes